CLINICAL TRIAL: NCT01387139
Title: Comparison of Ketamine Versus Co-Administration of Ketamine and Propofol for Procedural Sedation in a Pediatric Emergency Department
Brief Title: Ketamine Versus Co-administration of Ketamine and Propofol for Procedural Sedation in a Pediatric Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0835
Record Dates: First submitted 2011-05-20; First posted 2011-07-04 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Procedural Sedation and Analgesia
Keywords: Ketamine; Propofol; Procedural Sedation and Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Alone (Active Comparator): 1.0 milligrams/kilogram (mg/kg) ketamine with additional doses of 0.5 mg/kg ketamine as needed (maximum single dose based on 100 kilogram (kg) person)
  Interventions: Drug: Ketamine
- Ketamine Co-Administered with Propofol (Experimental): 0.5 mg/kg ketamine and 0.5 mg/kg propofol with additional doses of 0.25 mg/kg ketamine and 0.25 mg/kg propofol as needed (maximum single dose based on 100 kg person)
  Interventions: Drug: Ketamine Co-administered with Propofol

INTERVENTIONS:
Drug: Ketamine — 1.0 milligrams/kilogram (mg/kg) ketamine with additional doses of 0.5 mg/kg ketamine as needed (maximum single dose based on 100 kilogram (kg) person)
  Arms: Ketamine Alone
Drug: Ketamine Co-administered with Propofol — 0.5 mg/kg ketamine and 0.5 mg/kg propofol with additional doses of 0.25 mg/kg ketamine and 0.25 mg/kg propofol as needed (maximum single dose based on 100 kg person)
  Arms: Ketamine Co-Administered with Propofol

SUMMARY:
The purpose of this study is to compare the effectiveness of the co-administration of intravenous ketamine and propofol to intravenous ketamine as a single agent for procedural sedation in the pediatric emergency department. The investigators hypothesize that patients receiving co-administration of ketamine and propofol will have a lower rate of adverse events, compared to patients receiving ketamine for procedural sedation.

DETAILED DESCRIPTION:
Procedural sedation and analgesia (PSA) is a frequent occurrence in pediatric emergency departments. The goals of PSA include maximizing analgesia and amnesia, and minimizing adverse events while ensuring stable cardiopulmonary function. For decades, ketamine has been the main pharmacologic agent used for pediatric PSA. Numerous studies support the use of ketamine for sedation, amnesia, and analgesia on children undergoing painful procedures in the emergency department setting. Research has continually shown ketamine to cause emergence phenomenon, laryngospasm and vomiting.

Propofol is a sedative-hypnotic widely used for procedural sedation in adult emergency departments. The advantages of propofol include rapid onset, with quick and predictable recovery time, and antiemetic effects. Disadvantages include dose-dependent hypotension, bradycardia, respiratory depression, as well as pain with injection. In addition, propofol does not provide any analgesia.

Ketamine and propofol administered together have been successfully utilized in a variety of settings, including dermatologic, cardiovascular, and interventional radiological procedures in children. The co-administration of ketamine and propofol has been shown to preserve sedation while minimizing the respective adverse events. When used in combination, doses administered of each can be reduced, while producing a more stable hemodynamic and respiratory profile. Furthermore, this combination may reduce the frequency of emergence reactions, vomiting, and the pain of propofol injection.

To date, there are no randomized controlled trials evaluating the co-administration of ketamine and propofol versus ketamine monotherapy for PSA in the Pediatric Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 3 years and < 21 years
* American Society of Anesthesiologists (ASA) class I or II
* Fracture or dislocation requiring reduction under procedural sedation with ketamine as deemed by the attending emergency medicine physician
* Parent/Legal Guardian or Patient (if 18 years of age or older) has already given verbal consent for procedural sedation as part of standard care for their condition

Exclusion Criteria:

* Hypertension (Blood Pressure > 95th percentile for age)
* Glaucoma or acute globe injury
* Increased intracranial pressure or central nervous system mass lesion
* Porphyria
* Previous allergic reaction to ketamine
* Previous allergic reaction to Propofol or its components including soybean oil, glycerol, egg lecithin, and disodium edentate
* Disorders of lipid metabolism including primary hyperlipoproteinemia, diabetic hyperlipemia, or pancreatitis
* Mitochondrial myopathies or disorders of electron transport
* Pregnancy
* Parent, guardian or patient unwilling/unable to provide informed consent/assent

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Bajaj, MD, MPH, Principal Investigator — University of Colorado, Denver; Keith Weisz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Background] Roback MG, Wathen JE, Bajaj L, Bothner JP. Adverse events associated with procedural sedation and analgesia in a pediatric emergency department: a comparison of common parenteral drugs. Acad Emerg Med. 2005 Jun;12(6):508-13. doi: 10.1197/j.aem.2004.12.009. PMID 15930401
- [Background] Wathen JE, Roback MG, Mackenzie T, Bothner JP. Does midazolam alter the clinical effects of intravenous ketamine sedation in children? A double-blind, randomized, controlled, emergency department trial. Ann Emerg Med. 2000 Dec;36(6):579-88. doi: 10.1067/mem.2000.111131. PMID 11097698
- [Background] Akin A, Esmaoglu A, Guler G, Demircioglu R, Narin N, Boyaci A. Propofol and propofol-ketamine in pediatric patients undergoing cardiac catheterization. Pediatr Cardiol. 2005 Sep-Oct;26(5):553-7. doi: 10.1007/s00246-004-0707-4. PMID 16132313
- [Background] Akin A, Esmaoglu A, Tosun Z, Gulcu N, Aydogan H, Boyaci A. Comparison of propofol with propofol-ketamine combination in pediatric patients undergoing auditory brainstem response testing. Int J Pediatr Otorhinolaryngol. 2005 Nov;69(11):1541-5. doi: 10.1016/j.ijporl.2005.04.011. Epub 2005 Jun 3. PMID 15936092
- [Background] Akin A, Guler G, Esmaoglu A, Bedirli N, Boyaci A. A comparison of fentanyl-propofol with a ketamine-propofol combination for sedation during endometrial biopsy. J Clin Anesth. 2005 May;17(3):187-90. doi: 10.1016/j.jclinane.2004.06.019. PMID 15896585
- [Background] Barbi E, Marchetti F, Gerarduzzi T, Neri E, Gagliardo A, Sarti A, Ventura A. Pretreatment with intravenous ketamine reduces propofol injection pain. Paediatr Anaesth. 2003 Nov;13(9):764-8. doi: 10.1046/j.1460-9592.2003.01150.x. PMID 14617116
- [Background] Sharieff GQ, Trocinski DR, Kanegaye JT, Fisher B, Harley JR. Ketamine-propofol combination sedation for fracture reduction in the pediatric emergency department. Pediatr Emerg Care. 2007 Dec;23(12):881-4. doi: 10.1097/pec.0b013e31815c9df6. PMID 18091596
- [Background] Willman EV, Andolfatto G. A prospective evaluation of "ketofol" (ketamine/propofol combination) for procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2007 Jan;49(1):23-30. doi: 10.1016/j.annemergmed.2006.08.002. Epub 2006 Oct 23. PMID 17059854
- [Background] Cravero JP, Beach ML, Blike GT, Gallagher SM, Hertzog JH; Pediatric Sedation Research Consortium. The incidence and nature of adverse events during pediatric sedation/anesthesia with propofol for procedures outside the operating room: a report from the Pediatric Sedation Research Consortium. Anesth Analg. 2009 Mar;108(3):795-804. doi: 10.1213/ane.0b013e31818fc334. PMID 19224786
- [Background] American Academy of Pediatrics; American Academy of Pediatric Dentistry; Cote CJ, Wilson S; Work Group on Sedation. Guidelines for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures: an update. Pediatrics. 2006 Dec;118(6):2587-602. doi: 10.1542/peds.2006-2780. PMID 17142550
- [Background] Bhatt M, Kennedy RM, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM, Roback MG; Consensus Panel on Sedation Research of Pediatric Emergency Research Canada (PERC) and the Pediatric Emergency Care Applied Research Network (PECARN). Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009 Apr;53(4):426-435.e4. doi: 10.1016/j.annemergmed.2008.09.030. Epub 2008 Nov 20. PMID 19026467
- [Background] Macnab AJ, Levine M, Glick N, Phillips N, Susak L, Elliott M. The Vancouver sedative recovery scale for children: validation and reliability of scoring based on videotaped instruction. Can J Anaesth. 1994 Oct;41(10):913-8. doi: 10.1007/BF03010934. PMID 8001210
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Started | 99 | 84
Completed | 99 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol | Total
Number analyzed (Participants) | 99 | 84 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 99 | 84 | 183
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 74 | 54 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 72 | 62 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 99 | 84 | 183

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: We will record all adverse events during the sedation, and then perform a follow-up call to determine if any additional adverse events occured after discharge.
Time Frame: From enrollment through completion of follow-up, up to 7 days
Population: Adverse events
Measure: Number; unit: participants
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
participants
  Respiratory depression | 12 | 15
  Cardiovascular event | 1 | 0
  vomiting/retching | 21 | 18
  Unpleasant recovery reaction | 4 | 2

2. Secondary Outcome: Recovery Time
Description: Time until the patient has a Vancouver Sedation Recovery Scale Score of 18 or greater.
Time Frame: Once Vancouver Sedation Recovery Scale Score reaches 18 or greater, on average less than 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
minutes | 44 [19 to 69] | 43.5 [17.5 to 67.5]

3. Secondary Outcome: Efficacy of Sedation
Description: Efficacy is defined as:
  1. The patient does not have unpleasant recall of the procedure.
  2. The patient did not experience sedation-related adverse events resulting in abandonment of the procedure or a permanent complication or an unplanned admission to the hospital or prolonged emergency department (ED) observation
  3. The patient did not actively resist or require physical restraint for completion of the procedure. The need for minimal redirection of movements should not be considered as active resistance or physical restraint.
  4. The procedure was successful
Time Frame: After procedure is completed, on average less than 1 hour
Measure: Number; unit: participants
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
participants | 97 | 81

4. Secondary Outcome: Parent Satisfaction
Description: Measured on a 10-point scale (1= least satisfied, 10= most satisfied)
Time Frame: After procedure is completed, on average less than 1 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale (1-10)
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
units on a scale (1-10) | 10 [9 to 10] | 10 [8 to 10]

5. Secondary Outcome: Physician Performing Procedure Satisfaction
Description: Measured on a 10-point scale (1= least satisfied, 10= most satisfied)
Time Frame: After procedure is completed, on average less than 1 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
units on a scale | 9 [7 to 10] | 8 [4 to 10]

6. Secondary Outcome: Nurse Satisfaction
Description: Measured on a 10-point scale (1= least satisfied, 10= most satisfied)
Time Frame: After procedure is completed, on average less than 1 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Number analyzed (Participants) | 99 | 84
units on a scale | 10 [8 to 10] | 8 [4 to 10]

ADVERSE EVENTS:
Arm/Group | Ketamine Alone | Ketamine Co-Administered With Propofol
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/84
Other Adverse Events (participants affected / at risk) | 38/99 | 33/84
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Alone (N=99) | Ketamine Co-Administered With Propofol (N=84)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 15 (15)
Vomiting (Gastrointestinal disorders) | 21 (21) | 18 (18)
Cardiovascular event (Cardiac disorders) | 1 (1) | 0 (0)
Unpleasant recovery Reaction (Psychiatric disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes